CLINICAL TRIAL: NCT02007811
Title: Prospective, Open-label, Multicentre Clinical Trial, Phase I/IIa, to Investigate the Safety and Tolerability of Allogeneic B-cell Concentrates CD3+-Depleted, CD19+-Enriched, Cryopreserved (Single Administration After Day 120 Following Allogeneic Stem Cell Transplantation (SCT), Donor-identical) in 4 Groups With Escalating Doses for Immune Response Enhancement, Measured as Response to a Antedated Single Vaccination
Brief Title: Open-label Clinical Trial to Investigate the Safety and Tolerability of Allogeneic B-cell Concentrates for Immune Reconstitution After Allogeneic Stem Cell Transplantation Measured as Response to a Antedated Single Vaccination
Acronym: B-cell therapy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: University Hospital Regensburg (Other); Wuerzburg University Hospital (Other); University Hospital, Essen (Other); German Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UKER-BLZ-PH1
Record Dates: First submitted 2013-11-21; First posted 2013-12-11 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Chronic Myeloid Leukemia; Non Hodgkin's Lymphoma; Hodgkin's Disease; Myelodysplastic Syndrome; Multiple Myeloma; Aplastic Anemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Lymphoma, Non-Hodgkin; Hodgkin Disease; Myelodysplastic Syndromes; Multiple Myeloma; Anemia, Aplastic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- allogeneic donor derived B-lymphocytes (Experimental)
  Interventions: Biological: allogeneic donor derived B-lymphocytes

INTERVENTIONS:
Biological: allogeneic donor derived B-lymphocytes — CD3+-depleted, CD19+-enriched, cryopreserved (single administration after day 120 following allogeneic stem cell transplantation, donor-identical) in 4 groups with escalating doses

SUMMARY:
The reconstitution of a functioning immune system after allogeneic stem cell transplantation takes months to years. Particularly memory B-lymphocytes reconstitute poorly with the current conditioning regimes. During the period of intense immune suppression the patients are extremely susceptible to bacterial, fungal and, most importantly, viral infections.The adoptive transfer of B-lymphocytes from the stem-cell donor might significantly enhance humoral immunity for the patient. Aim of the study is to evaluate a new cellular therapy with B-lymphocytes regarding safety. A booster vaccination after B-lymphocyte transfer will evaluate the functionality of the transferred B-lymphocytes in the patient.

ELIGIBILITY:
Inclusion Criteria:

1. patients after allogeneic stem cell transplantation
2. Serostatus for EBV: R-/D- oder R+/D- oder R+/D+

Exclusion Criteria:

1. Serostatus for EBV: R-/D+
2. Severe acute Graft versus Host Disease (GvHD) (Glucksberg grade III und IV)
3. Chronic GvHD in middle- or high-risk group according to NIH staging
4. Rituximab administration after SCT
5. >10.000 EBV DNA copies/ml plasma
6. Recurrence of the haematological disorder needing therapeutic intervention
7. Secondary transplantation
8. SCT with transplant from a haploidentical donor
9. SCT with transplant from umbilical cord blood
10. CD34+-enriched transplant
11. in vitro T-cell depleted transplant
12. Pregnant or breast-feeding female

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with EBV DNA copies/ml plasma higher than 50,000 | for 120 days after administration of study medication
Number of participants with signs of a post-transplant lymphoproliferative disorder (PTLD) | for 120 days after administration of study medication
Number of participants with adverse events (AEs), adverse reactions (ARs), serious adverse events (SAEs), serious adverse reactions (SARs) and suspected unexpected serious adverse reaction (SUSARs) | for 120 days after administration of study medication

SECONDARY OUTCOMES:
Change in the frequency of antibody-producing cells between dose groups | before and 7 days after preponed single vaccination
Change of mean absolute number of B-lymphocytes, naïve B-lymphocytes and memory B-lymphocytes between dose groups. | 1 day before and up to 120 days after administration of study medication
Change of antigen-specific antibody concentration in serum/plasma between dose groups | 1 day before and up to 120 days after administration of study medication
Change of Cytomegalovirus (CMV) DNA copies/ml plasma between dose groups | 1 day before and up to 120 days after administration of study medication
Number of patients with >5,000 CMV DNA copies/ml plasma or with signs of organ infestation by CMV between dose groups. | up to 120 days after administration of study medication

CONTACTS AND LOCATIONS:
Overall Officials: Julia Winkler, MD, Principal Investigator — University Hospital Erlangen
Locations (1):
- Medical Department 5, University Hospital Erlangen, Erlangen, Germany

REFERENCES:
- [Derived] Winkler J, Tittlbach H, Schneider A, Vasova I, Strobel J, Herold S, Maas S, Spriewald BM, Repp R, Kordelas L, Mach M, Wolff D, Edinger M, Mackensen A, Winkler TH. Adoptive transfer of donor B lymphocytes: a phase 1/2a study for patients after allogeneic stem cell transplantation. Blood Adv. 2024 May 28;8(10):2373-2383. doi: 10.1182/bloodadvances.2023012305. PMID 38467031